CLINICAL TRIAL: NCT05965115
Title: The China Monoclonal Gammopathy Screening Project in First-degree Relatives of Patients With Multiple Myeloma (CHAPERONE) --A Multicenter Observational Study
Brief Title: The China M-protein Screening Project in First-degree Relatives of Myeloma Patient - The CHAPERONE Study
Acronym: CHAPERONE
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Peng Liu, Head of Department of Hematology, Shanghai Zhongshan Hospital
Other Study IDs: CHAPERONE
Record Dates: First submitted 2023-06-30; First posted 2023-07-28 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance
Keywords: Monoclonal Gammopathy of Undetermined Significance; Multiple Myeloma; Early Tumor Screening
MeSH Terms: conditions — Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Sample of Blood — All participants will receive M-protein screening by serum electrophoresis. Individuals with detected M-protein will undergo further diagnostic tests to determine their accurate diagnosis. Patients with monoclonal gammopathy of undetermined significance (MGUS) would be carefully assessed and followed up.

SUMMARY:
The goal of the China Monoclonal Gammopathy Screening Project in First-degree Relatives of Patients With Multiple Myeloma (CHAPERONE) study is to assess the clinical significance of screening for monoclonal gammopathy (M-protein) in first-degree relatives of patients with multiple myeloma in China population, and establish a prospective cohort of individuals with monoclonal gammopathy of undetermined significance (MGUS), a precursor conditions to multiple myeloma. We will study these patients as a means to identify risk factors for progression to symptomatic multiple myeloma.

DETAILED DESCRIPTION:
The CHAPERONE study aims to assess the clinical significance of screening for monoclonal gammopathy in first-degree relatives of patients with multiple myeloma in China.

The main objectives it aims to answer are:

* Main research objectives: To study the prevalence of MGUS, the time of disease progression, and its influencing factors in first-degree relatives of multiple myeloma patients in China.
* Secondary study objective: To explore the clinical/genomic/epigenetic features, survival, and quality of life of MGUS patients in first-degree relatives of multiple myeloma patients in China.

All participants will receive M-protein screening by serum electrophoresis. Individuals with detected M-protein will undergo further diagnostic tests, and patients with MGUS will be carefully assessed and followed up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female over the age of 18;
2. First-degree relatives (including parents, children, and biological siblings) have multiple myeloma diagnosed by the International Myeloma Working Group (IMWG) Myeloma Diagnostic Criteria;
3. Understand the purpose and procedure of this trial and voluntarily participate in this screening study;
4. Participants should be willing and able to follow the study follow-up plan and other protocol requirements.

Exclusion Criteria:

Patients with a known diagnosis of plasma cell diseases, such as MGUS, smoldering myeloma (SMM), or multiple myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first-degree relatives of patients with multiple myeloma in the Chinese population.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2035-08 (Estimated)

PRIMARY OUTCOMES:
The prevalence of monoclonal gammopathy of undetermined significance (MGUS) in MM first-degree relatives | 2 Years
  The prevalence of MGUS in MM first-degree relatives: defined as the proportion of MGUS cases among the total population ( MM first-degree relatives) receiving M-protein screening
Time to progression (TTP) from MGUS to overt multiple myeloma | 10 Years
  The time interval between the first diagnosis of MGUS and the first recording of participants and the diagnosis of myeloma. For participants who did not record disease progression to myeloma, the last follow-up date was used as the cut-off date.

SECONDARY OUTCOMES:
Overall survival of MGUS patients | 10 Years
  The time interval between the first diagnosis of MGUS and the recording of death from any cause. For participants whose death is not recorded, the cut-off date is the most recent point at which it is known that the participant is still alive.
Quality of life (QoL) of MGUS patients | 10 Years
  QoL evaluation was performed using the Patient Self-Rating Scale (EORTC QLQ - C30) during the case screening period and at each follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Liu, PhD, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital，Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Li J, Wang Y, Liu P. The impact on early diagnosis and survival outcome of M-protein screening-driven diagnostic approach to multiple myeloma in China: a cohort study. J Cancer. 2019 Aug 27;10(20):4807-4813. doi: 10.7150/jca.32103. eCollection 2019. PMID 31598151